CLINICAL TRIAL: NCT03944421
Title: The Effects of Replacing Red and Processed Meat With Quorn on Markers of Gastrointestinal Health
Brief Title: The Effects of Replacing Red and Processed Meat With Quorn on Biomarkers of Gut Health
Acronym: MYCOMEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Quorn (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: NorthumbriaU001
Record Dates: First submitted 2019-03-05; First posted 2019-05-09 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2019-05

CONDITIONS: Colorectal Cancer
Keywords: Genotoxicity; DNA damage; Gut Microbiota; Metabolites
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Dyrk Kinases

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Red and Processed Meat (Experimental): 240 grams (raw weight) of red and processed meat every day for 2 weeks
  Interventions: Other: Red and Processed Meat
- Quorn (Experimental): 240 grams (uncooked weight) of Quorn every day for 2 weeks
  Interventions: Other: Quorn

INTERVENTIONS:
Other: Red and Processed Meat — Integration of 240 grams (raw weight) of red and processed meat into daily diet for 2 week period.
  Arms: Red and Processed Meat
Other: Quorn — Integration of 240 grams (uncooked weight) of Quorn into daily diet for 2 week period.
  Other Names: Quorn Food
  Arms: Quorn

SUMMARY:
This study will evaluate the effects of substituting red and processed meat in the diet with Quorn; a meat replacement product, on biomarkers of gut health. This will be a crossover design where participants will take part in 2 study periods where they will consume a diet containing red and processed meat during one of the study periods, whereas in the other study period, they will consume a diet containing Quorn.

DETAILED DESCRIPTION:
There is a strong association between a diet which is high in red and processed meat, while low in fibre, and the incidence of colorectal cancer. This study aims to evaluate the effects of replacing red and processed meat in the diet with an alternative meat product such as Quorn, on biomarkers of gut health that may be associated with colorectal cancer.

Quorn is a product which has a considerable fibre component; thus, the replacement of red and processed meat with Quorn, will not only reduce the amount of compounds implicated to have deleterious effects in the gastrointestinal tract (E.G. haem, nitroso compounds, heterocyclic amines), but will also increase the delivery of fibre into the gastrointestinal system, that may well have an overall positive impact on gut health.

In this study, the participants will consume 240 grams (raw weight) of either red and processed meat, or Quorn each day for a 2 week period, this will be followed by a 4 week period where they will return to their usual dietary habits; before swapping to consume the alternative food (red/processed meat or Quorn) for another 2 week period.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-50 years.
* Not been diagnosed with colorectal cancer, or adenomas.
* Habitual omnivorous dietary pattern.
* BMI ≥18-30 kg/m2.
* Blood HbA1c <58mmol/mol (<6.5%) (not diagnosed with diabetes)
* Fasting total cholesterol<7.8 mmol/l
* Triglycerides <2.3 mmol/l
* Normal liver function (assessed by measuring liver enzymes in the screening blood sample).
* Blood pressure lower than BP <140/90 mmHg.
* Not suffering any cardiovascular diseases/ heart diseases e.g. stroke in the past 12 months.
* Do not suffer from chronic gastrointestinal problems (e.g. Inflammatory Bowel Disease, Irritable Bowel Syndrome, coeliac disease)
* Do not take supplements or medication that effects gastrointestinal health
* Not participated in a pre-/probiotic or laxative trial within the previous 3 months.
* Not been prescribed and/or taken antibiotics in the previous 6 months.
* No history of alcohol misuse based on self-reported alcohol intake and measurement of liver enzymes in the screening blood sample.

Exclusion Criteria:

* Been diagnosed with colorectal cancer and/or colorectal adenomas.
* Been diagnosed with gastrointestinal disorders (e.g. Inflammatory bowel disease, irritable bowel syndrome, coeliac disease)
* Adherence to a dietary pattern which excludes foods from an animal origin.
* Abnormal blood biochemistry based on standard clinical cut- offs, as well as blood markers not fitting the inclusion criteria set.
* Have history of food intolerances/allergies (e.g. gluten or dairy) or intolerances (e.g. lactose).
* Taking, or unwilling to stop taking anti-oxidant supplements (e.g. vitamin C, vitamin E, Multivitamin tablets, polyphenol supplements)
* Received antibiotics in the previous 6 months.
* Have participated in similar dietary or prebiotic/probiotics study in the previous 3 months.
* Current smoker.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-01-29 (Actual)

PRIMARY OUTCOMES:
Genotoxic potential of Faecal extracts from volunteers consuming intervention diets rich in red and processed meat versus diets containing Quorn | 2 weeks- Change from baseline following two week intervention with meat versus Quorn consumption
  Changes in the DNA damage causing capacity of aqueous stool extracts, assessed against HT29 and Caco-2 cells using the Comet assay.

SECONDARY OUTCOMES:
Oxidative Damage | 2 weeks- Change from baseline following two week intervention with meat versus Quorn consumption
  Changes in the concentration of 8-Hydroxyguanosine levels in urine samples.
Endogenous Short Chain Fatty Acid Production | 2 weeks- Change from baseline following two week intervention with meat versus Quorn consumption
  Changes from baseline in the concentration of short chain fatty acids in stool samples, measures of propionate, acetate, butyrate valerate and isovalerate via Gas Chromatography.
Gut Microbial Composition | 2 weeks- Change from baseline following two week intervention with meat versus Quorn consumption
  Evaluation of post-intervention changes in the composition of the stool microbiota composition from baseline samples.
Endogenous Production of Para-Cresol | 2 weeks- Change from baseline following two week intervention with meat versus Quorn consumption
  Change in the concentration of the genotoxic metabolite para-cresol in urine samples
Changes in MicroRNA Expression | 2 weeks- Change from baseline following two week intervention with meat versus Quorn consumption
  Evaluation of change in the abundance of microRNAs in plasma separated from blood samples following the intervention.

OTHER OUTCOMES:
Blood Cholesterol | 2 weeks
  Changes in levels of cholesterol in blood samples
Blood Glucose | 2 weeks
  Changes in levels of glucose in blood samples (HbA1c)

CONTACTS AND LOCATIONS:
Overall Officials: daniel M commane, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available within 18 months of study completion
Access Criteria: Northumbria University has plans to acquire a data repository for sharing data in the near future.

REFERENCES:
- [Derived] Farsi DN, Gallegos JL, Finnigan TJA, Cheung W, Munoz JM, Commane DM. The effects of substituting red and processed meat for mycoprotein on biomarkers of cardiovascular risk in healthy volunteers: an analysis of secondary endpoints from Mycomeat. Eur J Nutr. 2023 Dec;62(8):3349-3359. doi: 10.1007/s00394-023-03238-1. Epub 2023 Aug 25. PMID 37624376
- [Derived] Farsi DN, Gallegos JL, Koutsidis G, Nelson A, Finnigan TJA, Cheung W, Munoz-Munoz JL, Commane DM. Substituting meat for mycoprotein reduces genotoxicity and increases the abundance of beneficial microbes in the gut: Mycomeat, a randomised crossover control trial. Eur J Nutr. 2023 Apr;62(3):1479-1492. doi: 10.1007/s00394-023-03088-x. Epub 2023 Jan 18. PMID 36651990